CLINICAL TRIAL: NCT01794598
Title: HF-ACTION Depression Education Substudy
Brief Title: Preliminary Study Examining Heart Failure Patients Responses to Depression Education
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 5132; 5132-03-8R0ER (Other: Duke legacy protocol ID)
Record Dates: First submitted 2012-02-17; First posted 2013-02-20 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Heart Failure
Keywords: Heart failure; depression; depression care education
MeSH Terms: conditions — Heart Failure; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational materials (Experimental): Receiving educational materials of depression care
  Interventions: Behavioral: Receiving educational material of depression care
- No educational materials (Sham Comparator): Receiving an envelope but no inclusion of educational materials of depression care
  Interventions: Behavioral: Receiving educational material of depression care

INTERVENTIONS:
Behavioral: Receiving educational material of depression care — The educational material provides patients about depression management

SUMMARY:
Purpose of the Study: The significant impact of depression on the poor prognosis and functional restrain, recognition and successful treatment of depression in patients with Chronic Heart Failure (CHF) may result in improvement of overall outcome of those patients. However, depression comorbid with CHF has been overlooked in the real practice. Therefore, the investigators are proposing a study to 1) assess the prognostic impact of depression in patients with stable CHF who have been managed as outpatients, and 2) assess whether provision of depression education to CHF patients will improve the care of depression.

Patients with chronic heart failure are enrolled into this study with a half of them are randomly assigned to receive a packet of depression education materials and then other half not. Participants and investigators both are blinded to the assignment. All the participants are provided a toll free phone number to contact the research team as needed. Depressive symptoms and patients knowledge of depression are assessed at baseline prior to randomization and at 1-month and 6-month following the enrollment.

Responses of the study participants, such as change of depressive symptoms, and requests for psychiatric help are examined between two groups.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

* LVEF ≤ 35%.
* NYHA class II, III, or IV heart failure for the previous three months despite a minimum of 6 weeks of treatment.
* Must be on optimal heart failure therapy according to AHA/ACC and HFSA heart failure guidelines, including treatment with ACEI and beta-blocker therapy, or have documented rationale for variation, including intolerance, contraindication, patient preference, or personal physician's judgment.

Exclusion Criteria:

* Age less than 18.
* Currently pregnant or intending to become pregnant in the next year.
* Cardiovascular procedure or hospitalization for any reason planned in the next 6 months.
* Expectation of receiving a cardiac transplant in the next six months.
* Unable to provide the study consent.
* Participation another clinical trial(s) that may interfere with follow-up or data collection for this study, or that may affect cardiovascular mortality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2004-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in recognition of study participant to depression care | Baseline, 1 month and 6 months
  To assess whether the provision of depression education materials will increase knowledge of the impact depression has on Congestive Heart Failure patients. This will be measured through study participants completion of a questionnaire to record their views on depression and depression care in a non-psychiatric setting.

SECONDARY OUTCOMES:
Change in response of study participant to depression care | Baseline, 1 month, and 6 months
  Response of participants to depression care was measured by use of the Beck Depression Inventory scale (BDI), PHQ-9 (the 9 items of the depression scale of the Patient Health Questionnaire) and an anxiety questionnaire and a toll-free contact number to access free psychiatric consultants at the coordinating center. A contact log was kept documenting subject ID, reason for call, number of contacts and duration of the call.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jiang, MD, Principal Investigator — Duke University